CLINICAL TRIAL: NCT06674967
Title: Efficacy and Safety of Left Bundle Area Pacing Vs Right Ventricular Apical Pacing in Patients with Atrioventricular Block
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Karim Mohamed Eltaher Abdelrahman Aly, Assistant lecturer, Assiut University
Other Study IDs: LBB pacing vs RV pacing in AVB
Record Dates: First submitted 2024-10-14; First posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Atrio-Ventricular Block
Keywords: Efficacy; Safety; RV apical pacing; LBB area pacing; Atrioventricular block
MeSH Terms: conditions — Atrioventricular Block

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — venous blood sample for routine investigations as in complete blood count
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- LBB area pacing group: study group with LBB area pacing
- RV apical pacing area: study group with RV apical pacing

SUMMARY:
This study will address whether LBBaP is superior to RVAP in terms of safety and efficacy

DETAILED DESCRIPTION:
* Cardiac pacing is an effective therapy for treating patients with bradycardia due to sinus node dysfunction or atrioventricular block. However, traditional right ventricular apical pacing (RVAP) causes electric and mechanical desynchrony, increasing the risk for atrial arrhythmias and heart failure.
* .Cardiac resynchronization therapy(CRT)is another pacing modality employed for treatment of HF .Clinical studies have demonstrated that CRT promotes left ventricular reverse remodelling and reduces morbidity and mortality in patients with HF . Although CRT's benefits are well demonstrated, the therapy has been associated with significantly high non-response rate(30-40%).Also, the BVP is a non-physiological approach that requires two leads to activate the ventricular myocardium and not the specialized conduction system
* Therefore, there is a need to develop a physiological pacing approach that provides synchronized contraction of the ventricles
* Although His bundle pacing (HBP)has been widely used as a physiological pacing modality, it is limited by challenging implantation technique, unsatisfactory success rate in patients with wide QRS wave, high pacing capture threshold, and early battery depletion.
* Recently, the left bundle branch pacing (LBBP), defined as the capture of the left bundle branch (LBB) via trans ventricular septal approach, has emerged as a new physiological pacing modality.
* this approach has been found to provide physiological pacing that guarantees electrical synchrony of the left ventricle with a low pacing threshold.
* LBBP implantation is done by The Select Secure lead (model 3830) and Select Site C315HisorC304His sheaths are used in operation, while an electrophysiological multichannel recorder is used to simultaneously document intracardiac EGMs and 12-lead ECG .the Pacing System Analyzer (PSA) is used to test the pacing parameters and record intracardiac EGMs. The operation process can be summarized as follows: (1) establishment of the venous access and determination of the initial LBBP site; (2) introducing a pacing lead into the right ventricle and screwing it into the interventricular septum(IVS) until it reached in the LBB areas;(3) assessing the lead depth into ventricular septum and confirming LBB capture; (4)removing the sheath and providing the slack; and(5)programming the pulse generator.
* There is a limited number of clinical studies, featuring small sample sizes, that have shown that, compared with right ventricular apex pacing (RVAP), the QRS duration of postoperative ECG in LBBaP patients is narrower and the cardiac systolic function is improved. Also, there have been limited number of randomized controlled trials (RCTs) evaluating the efficacy and safety of LBBaP in patients with atrioventricular block (AVB) versus those with RVAP.

ELIGIBILITY:
Inclusion Criteria :

* Patients with AVB who meet indications for pacemaker
* Implantation with an estimated percentage of ventricular pacing ≥50%
* Ability to provide informed consent

Exclusion Criteria:

* Failure to cooperate with follow-up.
* Persistent atrial fibrillation.
* Patients with heart failure (LVEF) ≤35%,
* Estimated glomerular filtration rate less than 30 ml/min.
* Septic shock
* advanced malignant tumor.
* Pregnancy or prepared to get pregnant
* Cardiac tamponade or major hemopericardium

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: . Patients with AVB who meet indications for pacemaker , with an estimated percentage of ventricular pacing ≥50%
Sampling Method: Non-Probability Sample
Enrollment: 42 (Estimated)
Dates: Start 2024-11-30 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
effectiveness with LBB pacing | 3 years
  Assess left ventricular global strain using speckle tracking echocardiography (percentage)
Incidence of adverse events in patient with LBB pacing | 3 years
  Malignant arrhythmia(Yes/No)
Incidence of septal perforation | 3 years
  Detect septal perforation(Yes/No)

SECONDARY OUTCOMES:
Major Adverse Cardiovascular Events | 3 years
  • All-cause mortality (Yes or No) cardiovascular deaths (Yes or No) rehospitalisation with heart failure (Yes or No) Lead dislocation (Yes or No) Lead infection. (Yes or No)

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, Asyut, Asyut Governorate, Egypt